CLINICAL TRIAL: NCT04176926
Title: Validation of Software for Assessment of Atrial Fibrillation From Data Acquired by a Wearable Smartwatch
Status: Completed | Type: Observational
Sponsor: Fitbit LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 129-0360-01
Record Dates: First submitted 2019-11-21; First posted 2019-11-25 (Actual); Last update posted 2020-04-09 (Actual); Status verified 2020-04

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Electrocardiography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: SR: Group 1: Subjects in the sinus rhythm (SR) cohort should not have any history of atrial fibrillation and should not be in atrial fibrillation or other atrial arrhythmia at the time of enrollment based on the screening ECG.
  Interventions: Diagnostic Test: Electrocardiogram
- Group 2: AF: Group 2: Subjects in the atrial fibrillation (AF) cohort must have a known history of AF and must be in AF at the time of enrollment based on the screening ECG.
  Interventions: Diagnostic Test: Electrocardiogram

INTERVENTIONS:
Diagnostic Test: Electrocardiogram — Diagnostic Test: Simultaneous assessment of heart rhythm by 12-lead ECG and wearable device characterization of heart rhythm.

SUMMARY:
The goal of this study is to validate the Fitbit ECG software algorithm's ability to detect atrial fibrillation using data derived from a Fitbit wrist-worn consumer device that features a single lead ECG. The performance of the software application will be measured against centralized Core Lab physician-adjudicated 12-lead ECG tracings from FDA cleared ECG monitors as reference standards. The Fitbit software is intended as a pre-screening technology. It should identify candidates who may benefit from further evaluation. The software is not intended to be a diagnostic system.

ELIGIBILITY:
Inclusion Criteria:

* Women and men 22 years of age or older
* Capable of giving informed consent
* Sufficient manual dexterity to capture an ECG from the Fitbit wrist-worn device.
* Subjects in the atrial fibrillation (AF) cohort must have a known history of AF and must be in -AF at the time of enrollment based on the screening ECG

Exclusion Criteria:

* Anti-arrhythmic (rhythm control) medication use (such as amiodarone or flecainide)
* Cardiac pacemaker or implantable cardioverter-defibrillator
* History of a life-threatening rhythm such as ventricular tachycardia or ventricular fibrillation
* Subjects in the sinus rhythm (SR) cohort should not have any history of atrial fibrillation and should not be in atrial fibrillation or other atrial arrhythmia at the time of enrollment based on the screening ECG

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited at the individual clinical sites. Subjects may be recruited during routine clinic visits or may be asked to come in specifically for this study.
Sampling Method: Non-Probability Sample
Enrollment: 472 (Actual)
Dates: Start 2019-10-29 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2020-03-02 (Actual)

PRIMARY OUTCOMES:
Evaluate the software algorithm's ability to classify a heart rhythm as sinus rhythm or atrial fibrillation from a waveform equivalent to a Lead I ECG. | Through study completion, an average of 4 months
  Sensitivity and specificity of the software algorithm in classifying sinus rhythm and atrial fibrillation from the equivalent of a Lead I ECG waveform, compared with physician's interpretation of a standard 12-lead ECG. Performance goals are 90% (sensitivity) and 92% (specificity)

SECONDARY OUTCOMES:
Confirm the software's ability to produce a waveform clinically equivalent to a Lead I ECG from a clinical reference device (12-lead ECG). | Through study completion, an average of 4 months
  Qualitative assessment of the software produced waveform to reference Lead I from 12-lead ECG. Goal is >0.80 of strips appear to overlay to the unaided eye.
  Comparison of R-wave amplitudes between the Fitbit waveform and the clinical reference. Goal is >0.80 of R-wave amplitudes to be within 2mm.

CONTACTS AND LOCATIONS:
Overall Officials: Venkatesh Raman, MD, Principal Investigator — Medstar Health Research Institute
Locations (10):
- United States (9):
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Bioclinica Research Orlando, Orlando, Florida
  - Bioclinica Research The Villages, The Villages, Florida
  - PMG Research of Dupage, Winfield, Illinois
  - PMG Research of McFarland, Ames, Iowa
  - PMG Research of Rocky Mount, Rocky Mount, North Carolina
  - PMG Research of Piedmont Healthcare, Statesville, North Carolina
  - PMG Research of Wilmington, Wilmington, North Carolina
  - PMG Research of Charleston, Mt. Pleasant, South Carolina
- Onassis Cardiac Surgery Center, Kallithea, Greece

IPD SHARING:
Plan to Share IPD: No